CLINICAL TRIAL: NCT06211803
Title: Clinical Application of the Prototype J-PET Device
Acronym: JPETClinic
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Ewa Stępień, PhD, Head of Department of Medical Physics, Jagiellonian University
Other Study IDs: KB16/2022; TEAM POIR.04.04.00-00-4204/17 (Other Grant/Funding Number: Foundation for Polish Science); 2021/42/A/ST2/00423 (Other Grant/Funding Number: National Science Centre of Poland); 2021/43/B/ST2/02150; (Other Grant/Funding Number: National Science Centre of Poland); SPUB/SP/490528/2021 (Other Grant/Funding Number: Ministry of Education and Science of Poland); CRP/0641.221.2020 (Other Grant/Funding Number: Jagiellonian University)
Record Dates: First submitted 2023-12-28; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Neurodegenerative Diseases; Brain Neoplasms; Neuroendocrine Tumors
Keywords: PSMA; PET; FDG; DOTATATE; positronium; Somatostatin analogues
MeSH Terms: conditions — Neurodegenerative Diseases; Brain Neoplasms; Neuroendocrine Tumors | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- J-PET group: The patient is referred for a PET/CT scan, in accordance with recognized indications for examining the brain or the entire body.
  Interventions: Diagnostic Test: Positron-Emission Tomography Imaging

INTERVENTIONS:
Diagnostic Test: Positron-Emission Tomography Imaging — Examination of radiation distribution in the patient brain and body after completing a routine examination on a PET diagnostic device. J-PET prototype tests will be carried out in patients who have undergone a classic PET examination after administration of [18F]FDG), [68Ga]Ga-PSMA or [68Ga]Ga-DOTATATE). The duration of the additional exam will be approximately 20 minutes.
  Other Names: PET Imaging; PET Scan; Positron-Emission Tomography

SUMMARY:
Positron emission tomography (PET) is a diagnostic imaging technique that uses positron emission (e-) to image changes in diagnosed tissues. Detector systems are an important part of PET scanners. They can convert gamma photons into fluorescent photons to obtain information about energy, time and position, of the gamma photons obtained through the use of an appropriate positron-emitting radiopharmaceutical. Conventional PET scanners are expensive mostly because they require the use of LSO (lutetium oxyorthosilicate) or LYSO (lutetium yttrium oxyorthosilicate) scintillation crystals. Such crystal scintillators are very costly and difficult to obtain, which limits accessibility of the PET- scanners. The prototype J-PET scanner tested in this trial uses plastic scintillators in which different physical phenomena occur compared to crystal scintillators. In addition, the J-PET scanner prototype is equipped with unique software enabling three-photon imaging, based on the annihilation resulting from the formation of the orto-positronium (o-Ps) in diagnosed tissue. The aim of this study is to demonstrate the clinical acceptability of such scanners based on plastic scintillators, which can additionally collect and process information on the lifetime of o-Ps derived from routinely used radiopharmaceuticals. Additionally, the aim of this study is to demonstrate the use of the new diagnostic indicator "positronium biomarker" in a prospective study, compared to routine diagnostic scanning.

DETAILED DESCRIPTION:
The J-PET scanner is the world's first positron tomograph based on plastic strip scintillators to measure the lifetime of the ortho-positronium (o-Ps) atom. This is a modular scanner, designed and installed at the Department of Experimental Particle Physics and Applications of the Jagiellonian University in Krakow. The J-PET scanner is based on technology patented in 2014 and 2016.

The J-PET scanner, unlike PET scanners commonly used in diagnostics, has three important features:

1. J-PET scintillators are made of plastic instead of expensive-to-produce LSO (lutetium oxyorthosilicate) or LYSO (lutetium yttrium oxyorthosilicate) scintillation crystals use in regular PET scanners;
2. J-PET is modular and can be adapted to the patient's size and expanded to a total-body PET scanner because;
3. J-PET can be used to test an additional parameter called the "positronium biomarker" which has not been used so far.

Ad. 1. Conventional PET scanners use LSO or LYSO scintillation crystals, which exploit the photoelectric effect and convert gamma photons into fluorescent photons to obtain information on the energy, time and position of gamma photons emitted by the positron annihilation (e+) process obtained by using an appropriate e+ emitting radiopharmaceutical. In plastic scintillators used in J-PET, the Compton effect is used, i.e. the phenomenon of scattering of high-energy photons on free or weakly bound electrons of the scintillator.

Ad. 2. The modular J-PET scanner can also be easily integrated with existing computed tomography (CT) systems, allowing for simultaneous conduction of both types of examinations.

Ad. 3. Positronium imaging is applied in the J-PET scanner. The PET technique uses radioisotopes that emit positron radiation (beta+). Traditional PET scanners image the distribution of gamma ray photons produced by the annihilation of an electron (e-) and a positron (e+). Annihilation may be preceded by the appearance of a positron atom - a quasi-stable system composed of an electron (e-) and its antiparticle - positron (e+), which occurs in approximately 30-40% of all annihilations occurring in the patient's body.

The time of such annihilation taking place through the state of the positronium atom depends on whether a positronium will be created in which e- and e+ will have parallel spins (triplet state ↑↑, this system is called ortho-positronium - o-Ps) or antiparallel spins (state singlet ↑ ↓, this system is called para-positronium - p-Ps). The average life time of o-Ps in vacuum is more then 1000 times longer (142 nano-seconds [ns]), then the average life time of p-Ps (125 pico-seconds [ps]). The average lifetime of o-Ps in a vacuum is over 1000 times longer (142 nanoseconds [ns]) than the average lifetime of p-Ps (125 picoseconds [ps]). The second difference is that o-Ps annihilation takes place over 3 photons, which has not been detected so far and which traditional PET. the annihilation time of the o-Ps atom can be an additional diagnostic parameter ("positronium biomarker") to be measured and analyzed in the J-PET scanner.

The clinical application of such "positronium biomarker" in terms of lesion detection, image quality and quantification is yet to be determined, which this study aims to address.

ELIGIBILITY:
Inclusion Criteria:

The patient is referred for a PET/CT scan, in accordance with recognized indications for examining the brain or the entire body.

* Age over 18 years
* Informed, voluntary consent to participate in the study

Exclusion Criteria:

* Pregnant women, breastfeeding women
* People with a previously diagnosed allergy to radiopharmaceuticals
* age under 18 years
* Lack of cooperation with the patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The research group in this study consisted of patients who were diagnosed at the Department of Nuclear Medicine of the Medical University of Warsaw. Patients underwent routine diagnostic positron emission tomography (PET) examination to diagnose diseases of the central nervous system (CNS).
  Patient characteristics:
  Patients were over 18 years of age. They were of Polish origin, white.
  The patients represented a variety of CNS disorders, including:
  Brain tumors, such as glial tumors, solid tumors and primary tumors of the nervous system, Neurodegenerative diseases, Neuroendocrine tumors.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Assessment of the quality of tests performed using J-PET prototype | Initial analyzes will last 12 weeks
  The reference result for the J-PET test will be the result obtained using a PET/CT device owned by the Department of Nuclear Medicine of the Medical University of Warsaw. For this purpose, the test images obtained with the two cameras will be analyzed by a team of medical physicists (phantom tests) and doctors, according to the principles given above.

SECONDARY OUTCOMES:
Analysis of positronium duration in the disease focus and reference area | It is planned that the first results will be obtained after 6 months.
  The lifetime of positronium is a parameter characterizing the examined structures, including the structures of brain tissues. The J-PET group proposed the use of positronium lifetime as a new diagnostic biomarker. There are currently no similar studies in the literature.

CONTACTS AND LOCATIONS:
Overall Officials: Leszek Krolicki, MD, PhD, Study Chair — Medical University of Warsaw; Ewa L Stepien, PhD, Study Director — Jagiellonian University; Pawel Moskal, PhD, Principal Investigator — Jagiellonian University
Locations (1):
- Department of Nuclear Medicine, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moskal P, Dulski K, Chug N, Curceanu C, Czerwinski E, Dadgar M, Gajewski J, Gajos A, Grudzien G, Hiesmayr BC, Kacprzak K, Kaplon L, Karimi H, Klimaszewski K, Korcyl G, Kowalski P, Kozik T, Krawczyk N, Krzemien W, Kubicz E, Malczak P, Niedzwiecki S, Pawlik-Niedzwiecka M, Pedziwiatr M, Raczynski L, Raj J, Rucinski A, Sharma S, Shivani, Shopa RY, Silarski M, Skurzok M, Stepien EL, Szczepanek M, Tayefi F, Wislicki W. Positronium imaging with the novel multiphoton PET scanner. Sci Adv. 2021 Oct 15;7(42):eabh4394. doi: 10.1126/sciadv.abh4394. Epub 2021 Oct 13. PMID 34644101
- [Background] Moskal P, Stepien EL. Prospects and Clinical Perspectives of Total-Body PET Imaging Using Plastic Scintillators. PET Clin. 2020 Oct;15(4):439-452. doi: 10.1016/j.cpet.2020.06.009. Epub 2020 Jul 29. PMID 32739047
- [Background] Moskal P, Kubicz E, Grudzien G, Czerwinski E, Dulski K, Leszczynski B, Niedzwiecki S, Stepien EL. Developing a novel positronium biomarker for cardiac myxoma imaging. EJNMMI Phys. 2023 Mar 24;10(1):22. doi: 10.1186/s40658-023-00543-w. PMID 36959477
- [Background] Dadgar M, Parzych S, Baran J, Chug N, Curceanu C, Czerwinski E, Dulski K, Elyan K, Gajos A, Hiesmayr BC, Kaplon L, Klimaszewski K, Konieczka P, Korcyl G, Kozik T, Krzemien W, Kumar D, Niedzwiecki S, Panek D, Perez Del Rio E, Raczynski L, Sharma S, Shivani S, Shopa RY, Skurzok M, Stepien EL, Tayefi Ardebili F, Tayefi Ardebili K, Vandenberghe S, Wislicki W, Moskal P. Comparative studies of the sensitivities of sparse and full geometries of Total-Body PET scanners built from crystals and plastic scintillators. EJNMMI Phys. 2023 Oct 11;10(1):62. doi: 10.1186/s40658-023-00572-5. PMID 37819578
- [Background] Moskal P, Kisielewska D, Curceanu C, Czerwinski E, Dulski K, Gajos A, Gorgol M, Hiesmayr B, Jasinska B, Kacprzak K, Kaplon L, Korcyl G, Kowalski P, Krzemien W, Kozik T, Kubicz E, Mohammed M, Niedzwiecki S, Palka M, Pawlik-Niedzwiecka M, Raczynski L, Raj J, Sharma S, Shivani, Shopa RY, Silarski M, Skurzok M, Stepien E, Wislicki W, Zgardzinska B. Feasibility study of the positronium imaging with the J-PET tomograph. Phys Med Biol. 2019 Mar 7;64(5):055017. doi: 10.1088/1361-6560/aafe20. PMID 30641509
- See also: Patent US8859973B2: Strip device and method for determining the location and time of reaction of the gamma quanta and the use of the device to determine the location and time of reaction of the gamma quanta in positron emission tomography — https://patents.google.com/patent/US8859973B2/en?oq=US+8%2c859%2c973